CLINICAL TRIAL: NCT05781035
Title: Moderate Sedation by Dexmedetomidine Versus General Anesthesia on the Diagnostic Yield of Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration: A Randomized Controlled Study
Brief Title: Dexmedetomidine Versus General Anesthesia on the Diagnosis of Endobronchial US-Guided Transbronchial Needle Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35719\9\22
Record Dates: First submitted 2023-02-23; First posted 2023-03-23 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Sedation; Dexmedetomidine; EBUS Guided Transbronchial Needle Aspiration
MeSH Terms: interventions — Dexmedetomidine; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine group (Active Comparator)
  Interventions: Procedure: dexmedetomidine
- general anesthesia group (Active Comparator)
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: dexmedetomidine — patients will recieve moderate sedation by dexmedetomidine as study group
  Arms: dexmedetomidine group
Procedure: general anesthesia — general anesthesia with neuromuscular blockade under controlled ventilation as control group.
  Arms: general anesthesia group

SUMMARY:
The aim of this study is to compare dexmedetomidine as moderate sedation versus general anathesia on the diagnostic yield of Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration

DETAILED DESCRIPTION:
Endobronchial ultrasound (EBUS)-guided transbronchial needle aspiration (EBUS-TBNA) has emerged as a highly effective, minimally invasive technique for sampling peribronchial, mediastinal, and lung masses for pathologic examination with low rate of complications, and costs.

Dexmedetomidine, is a high-affinity adrenergic agonist of the alpha 2 receptor, is a potential alternative sedative.

The use of dexmedetomidine does not lead to respiratory depression, or to a decline in cognitive skills or patient cooperation. This is because dexmedetomidine acts on the alpha-2 receptors in the locus coeruleus, in contrast to other sedatives (midazolam and propofol) which act on GABA receptors/cerebral cortex.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification II or III a requiring EBUS-TBNA based on suspicion of either benign or malignant disease in mediastinal or hilar lymph nodes (LNs) or masses or requiring EBUS-TBNA for mediastinal staging of lung cancer.

Exclusion Criteria:

* Suspected need for additional procedures other than EBUS-TBNA during planned bronchoscopy (e.g., need for navigational bronchoscopy, endobronchial biopsies, and therapeutic bronchoscopy)
* body mass index > 35 kg/m2
* allergies to any of the involved sedatives or anesthetic agents
* comorbidities contraindicating the EBUS procedure
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of Endobronchial ultrasound -guided transbronchial needle aspiration | During procedure
  The number of subjects in whom Endobronchial ultrasound -guided transbronchial needle aspiration provided a specific diagnosis will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Torky, Principal Investigator — Lecturer of Chest Department , Faculty of Medicine, Tanta University
Locations (1):
- Mohammad Fouad Algyar, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be provided under a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study